CLINICAL TRIAL: NCT03614273
Title: Nebulized Hypertonic Saline (3%) Versus Nebulized Adrenaline for Treatment of Bronchiolitis: A Randomized Control Trial
Brief Title: Nebulized Hypertonic Saline (3%) Versus Nebulized Adrenaline for Treatment of Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maulana Azad Medical College (Other)
Responsible Party: Principal Investigator, Jerin C Sekhar, Senior Resident, Department of Pediatrics, Maulana Azad Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: bronchiolitisjer90
Record Dates: First submitted 2018-07-13; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Bronchiolitis
Keywords: nebulization; adrenaline; hypertonic saline; bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — Saline Solution, Hypertonic; Epinephrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (HS) (Active Comparator): Nebulized with 4 ml of 3% hypertonic saline for a duration of 20 minutes
  Interventions: Drug: Hypertonic saline
- Group 2 (Adr) (Active Comparator): Nebulized with 0.1 mg/kg of adrenaline (non-racemic solution, 1:1000 concentration), which was diluted in normal saline to make it a 4 ml solution, for a duration of 20 minutes
  Interventions: Drug: Adrenaline

INTERVENTIONS:
Drug: Hypertonic saline — The nebulizations were administered via an oxygen run jet nebulizer, with a flow of 6-7 litres/min.
  Arms: Group 1 (HS)
Drug: Adrenaline — The nebulizations were administered via an oxygen run jet nebulizer, with a flow of 6-7 litres/min.
  Other Names: Epinephrine
  Arms: Group 2 (Adr)

SUMMARY:
The primary objective of this study was to compare the effectiveness of nebulized hypertonic saline (3%) and nebulized adrenaline in bronchiolitis. The secondary objective was to assess whether non-responders to initial therapy benefit from continuation of the same therapy.

This trial was conducted at a tertiary care teaching hospital over a period of one year in children with bronchiolitis presenting to the out-patient department and emergency. After obtaining a signed informed consent from the parents, all eligible children were assessed for baseline characteristics. A complete hemogram, chest X-ray were done in all and arterial blood gas analysis where ever required.

Computer generated random numbers were used for enrolment in consecutive manner and patients were randomly assigned into two groups. The first group received one dose (4ml) of nebulized hypertonic saline (3%).The second group received one dose (0.1 mg/kg) of nebulized adrenaline diluted in normal saline to make it a 4ml solution. Supportive care (nasal clearing, antipyretics, oxygenation, intravenous fluids) was done in both groups as necessary.

All children were reassessed 20 minutes after one dose of nebulization using the clinical score and a child was labelled as a "responder" if he showed an improvement in the clinical severity score by atleast 3 points after 20 minutes of nebulization. Both responders and non-responders were given a repeat dose of nebulization according to the group to which the child had been randomized, if: a) Severe audible wheeze with severe respiratory distress (severity score ≥9) b) Inability to maintain saturation >92% even on an O2 flow of 4 L/min. Non responders were given a maximum of three continuous doses of nebulization.

Child was considered fit for discharge if he/she was feeding well orally, there was no need for intravenous fluids, clinical severity score ≤3 and maintaining oxygen saturation >92% on room air for a period of more than 12 hours.

ELIGIBILITY:
Inclusion Criteria:

• Children aged 1 month to 2 years with moderate to severe bronchiolitis as per Wang score

Exclusion Criteria:

* Comorbidities such as congenital heart disease, bronchopulmonary dysplasia, cystic fibrosis, neurological diseases
* Known or suspected immunodeficiency
* Congenital malformations
* History of use of steroids within one week prior to presentation
* Severe disease requiring admission to intensive care unit/mechanical ventilation

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
Duration of hospital stay | During hospitalization, approximately 2 days
  Duration from the time of enrolment to the point at which the discharge criteria (feeding well orally, no need for intravenous fluids, clinical severity score ≤ 3 and maintaining oxygen saturation >92% on room air for a period of more than 12 hours) are met.

SECONDARY OUTCOMES:
Initial change in the Wang bronchiolitis clinical severity score | 20 minutes after the first nebulization
  A decrease in the Wang bronchiolitis clinical severity score by at least 3 points after 20 minutes of nebulization was considered as an improvement in the clinical condition. The Wang score ranges from 0 - 12 [0-4: mild, 5-8: moderate, 9-12: severe].
Number of hours of intravenous fluid requirement | During hospitalization, approximately 2 days
  Intravenous fluids were given to children unable to accept orally.
Number of hours of oxygen requirement | Till the time the child maintained a saturation of more than 94% for at least 4 hours
  Oxygen was administered when the saturation was less than 92%
Number of doses of nebulization needed | During hospitalization, approximately 2 days
  Indications for repeat dose were if:
  1. The child had severe audible wheeze with severe respiratory distress (severity score ≥9)
  2. The child was not able to maintain saturation >92% even on an oxygen flow of 4 L/min
Response after each nebulization | Assessed 20 minutes after each nebulization
  An improvement in the clinical severity score by at least 3 points after each nebulization.

CONTACTS AND LOCATIONS:
Overall Officials: Jerin C Sekhar, MD, Principal Investigator — Maulana Azad Medical College
Locations (1):
- Maulana Azad Medical College, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided